CLINICAL TRIAL: NCT00969735
Title: Cryoenergy Or Radiofrequency for Pulmonary Vein Isolation (COR Trial)
Brief Title: Cryoenergy Or Radiofrequency for Pulmonary Vein Isolation
Acronym: COR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Spanish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Nicasio Perez Castellano, MD, PhD, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COR-1
Record Dates: First submitted 2009-08-28; First posted 2009-09-01 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Catheter ablation; Cryoenergy; Implantable loop recorder; Pulmonary vein
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cryoablation (Active Comparator): Deflectable over-the-wire cryoablation balloon catheter (Arctic Front®, Cryocath Technologies)
  Interventions: Device: Pulmonary vein cryoablation
- Radiofrequency ablation (Active Comparator): Open irrigation ablation catheter (Navistar® Thermo-cool®, Biosense Webster Inc).
  Interventions: Device: Pulmonary vein radiofrequency ablation

INTERVENTIONS:
Device: Pulmonary vein cryoablation — A deflectable over-the-wire cryoablation balloon catheter (Arctic Front®) will be inflated and be positioned at each PV antrum. Then, cryoenergy will be delivered for 300 seconds. During cryoablation of the right PVs, the right phrenic nerve integrity will be monitored by the observation of right hemi-diaphragm contractions in response to right phrenic nerve pacing at the superior vena cava. Once the 4 PVs are cryoablated, the Arctic Front® catheter will be replaced by a decapolar PV mapping circular catheter (Lasso®, Biosense Webster, Diamond Bar, California, EEUU) to evaluate PV conduction. A second cryoablation application may be delivered at each PV, if necessary. Crossover to RF ablation to complete PV isolation is discouraged.
  Other Names: Cryoenergy balloon catheter ablation
  Arms: Cryoablation
Device: Pulmonary vein radiofrequency ablation — Ablation approach is ostial electrical isolation of all PVs with simultaneous use of the CARTO® electroanatomic mapping system (Biosense Webster, Tirat-Ha-Carmel, Israel). PV isolation will be performed by delivering RF energy at ostial sites with earliest PV potentials. Flow rate during the RF applications will be set at 15 mL/min (baseline 2 mL/min). Temperature and power limits will be set at 45ºC and 35 W. It will be allowed a 5 W reduction in power limit setting for small PVs (angiographic supero-inferior diameter > 12 mm), and a 5 W increase in areas located away from the esophagus, and for focal applications at sites resistant to ablation or recurrent gaps. The end-point of ablation will be to achieve bidirectional PV conduction block.
  Other Names: Pulmonary vein isolation
  Arms: Radiofrequency ablation

SUMMARY:
This is a prospective single-center randomized trial comparing the efficacy and safety of PV cryoablation with the Arctic Front® catheter versus the standard PV isolation using radiofrequency irrigated tip catheters. The efficacy of both strategies will be evaluated from a clinical point of view and from the detection and quantification of AF episodes by means of the Reveal XT® implantable loop recorder.

DETAILED DESCRIPTION:
Pulmonary vein (PV) isolation using a radiofrequency catheter is the most widespread technique for atrial fibrillation (AF) ablation. These procedures are difficult and time-consuming, because they require precise catheter manipulation and multiple radiofrequency applications. Thus, alternative techniques are being investigated to simplify the procedure. Recently, a cryoenergy balloon catheter has been developed for PV isolation (Arctic Front®, Cryocath Technologies). When this catheter is deployed at the PV antrum, it can create a circumferential lesion around the PV ostium by delivering a single cryoenergy application.

An implantable loop recorder for AF detection has been made available (Reveal XT®, Medtronic). It may help taking clinical decisions regarding anticoagulant and antiarrhythmic therapy and, at the same time, it may be a powerful tool to evaluate the efficacy of different therapeutic strategies.

This is a prospective single-center randomized trial comparing the efficacy and safety of PV cryoablation with the Arctic Front® catheter vs. the standard PV isolation using radiofrequency irrigated tip catheters. The efficacy of both strategies will be evaluated from a clinical point of view and from the detection and quantification of AF episodes by means of the Reveal XT® implantable loop recorder.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic recurrent paroxysmal AF (>2 episodes in the last 6 months), and
* Refractory to one or more class I or III antiarrhythmic drugs, and
* PV anatomy consisting of 4 single PV, with the long diameter of the right superior PV ostium ≤ 20 mm.

Exclusion Criteria:

* Age: < 18 or > 75 year-old
* Prior AF ablation
* Pregnancy
* Concomitant acute illness
* Hyperthyroidism
* Moderate to severe valvular heart disease
* Prior cardiac surgery
* Left atrium > 50 mm (anteroposterior diameter, parasternal long-axis view)
* Intracardiac thrombus
* Contraindications for anticoagulant therapy
* Inability to be followed in our center for at least 1 year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients without AF recurrences longer than 2 minutes | At the 12th month from ablation (using a blanking period of 3 months following ablation)

SECONDARY OUTCOMES:
Time to first AF recurrence longer than 2 minutes | Within the first 12 months from ablation (using a blanking period of 3 months following ablation, and without the use of any blanking period)
Cumulative burden of AF (number of AF episodes longer than 2 minutes) | At the 12th month from ablation (using a blanking period of 3 months following ablation)
Cumulative burden of AF (percentage of time in AF) | At the 12th month from ablation (using a blanking period of 3 months following ablation)
Proportion of patients with episodes of regular atrial tachycardia or atrial flutter requiring treatment with drugs, electrical cardioversion or ablation. | Within the first 12 months from ablation
Quality of Life and symptom status | At the 12th month from ablation
Proportion of patients with procedure-related complications | Within the first 12 months from ablation
Procedure time (minutes elapsed from the first puncture of the femoral vein to the removal of the last catheter) | At the end of the ablation procedure
Ablation time (minutes elapsed from the onset of the first energy delivery to the end of the last energy delivery). | At the end of the ablation procedure
Fluoroscopy time (minutes of fluoroscopy used during the entire ablation procedure) | At the end of the ablation procedure
Proportion of pulmonary veins remaining isolated | At the end of the ablation procedure

CONTACTS AND LOCATIONS:
Overall Officials: Nicasio Pérez Castellano, MD, PhD, Principal Investigator — Unidad de Arritmias, Hospital Clínico San Carlos, Madrid, Spain
Locations (1):
- Unidad de Arritmias, Hospital Clínico San Carlos, Madrid, Madrid, Spain